CLINICAL TRIAL: NCT06701214
Title: Discovering Outcomes in Clonal Hematopoiesis: The Clonal Hematopoiesis and Inflammation in VasculaturE (CHIVE) Registry and Biorepository
Brief Title: The Clonal Hematopoiesis & Inflammation in Vasculature Registry and Biorepository
Acronym: CHIVE
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Alexander Bick, Assistant Professor Medicine, Division of Genetic Medicine, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICCHEM20123; NCI-2021-00704 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2024-04-18; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Clonal Hematopoiesis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood collection — Blood will be taken from participants already undergoing blood collection
Other: Saliva collection — Undergo saliva collection
Other: Bone marrow collection — Bone marrow will be taken from participants already undergoing bone marrow collection

SUMMARY:
This study will investigate the association between clonal hematopoiesis and other conditions. Clonal hematopoiesis (CH) refers to the mutations in a person's stem cells which commonly affect people as they get older. These mutations have notably been linked to increased risk of certain cancers as well as increased risk of heart disease.

DETAILED DESCRIPTION:
Objectives:

* To develop the CHIVE Registry with CH patients or patients with elevated risk for CH in order to better characterize associated clinical outcomes and co-morbidities in these populations
* To improve understanding of cardiovascular phenotypes and risk of patients with known Clonal Hematopoiesis of indeterminate potential (CHIP) or Clonal Cytopenias of undetermined significance (CCUS)
* To investigate prognostic significance of CH mutations for the development hematologic malignancies
* To generate a CHIVE Biorepository to acquire patient samples to study the natural history of CH, and to make available to CH investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patient greater than or equal to 18 years old at time of consent
* Able to provide informed consent
* Idiopathic cytopenia (ICUS) or idiopathic cytoses (elevated blood counts without disease or explanation); clonal cytopenia of undetermined significance (CCUS), clonal hematopoiesis of indeterminate potential (CHIP) or individuals at higher risk for clonal hematopoiesis (ex. patients with known diagnosis of solid tumors or cardiovascular disease)

Exclusion Criteria:

* Unable to provide consent
* Diagnosis of active hematologic malignancy. For example, a diagnosis of CMML, AML, MDS, MPN; History of hematologic malignancy is NOT exclusionary if in complete remission (e.g. previous myeloma or lymphoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults >/= 18 years old with a mutation known to cause clonal hematopoiesis or at a higher risk of having a clonal hematopoiesis mutation.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
CHIVE Registry | Up to approximately 120 months
  Aggregate data will be utilized to better understand the association between clonal hematopoiesis and other conditions
CHIVE Biorepository | Up to approximately 120 months
  Number of biological samples collected and stored (Blood, saliva, bone marrow) for future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bick, MD, PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided